CLINICAL TRIAL: NCT06851702
Title: Observational Study for the Evaluation of Immune-mediated Endocrinological Adverse Events in Patients With Hematological Malignancies and Subjected to Treatment With Immune-checkpoint Inhibitors
Acronym: Endemato
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Endemato
Record Dates: First submitted 2025-01-29; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-10

CONDITIONS: Hematological Malignancies
Keywords: immune-checkpoint inhibitors; endocrinological adverse events
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retrospective / prospective observational study of endocrinological adverse events in hematologic patients treated with immunological checkpoint inhibitors

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort

* patients aged> 18 years
* cyto-histological diagnosis of mature lymphoproliferative syndrome of B or T lymphocyte origin
* advanced stage of illness (relapsed or refractory)
* patients undergoing treatment with immune anticheckpoint antibodies.
* written informed consent

Prospective cohort

* patients aged> 18 years
* cyto-histological diagnosis of mature lymphoproliferative syndrome of B or T lymphocyte origin
* advanced stage of illness (relapsed or refractory)
* patients who are candidates for therapy with anticheckpoint immune antibodies (it is specified that this therapy is completely independent of the subject's participation in the study).
* written informed consent

Exclusion Criteria:

* Severe, acute and chronic medical or psychiatric disorders that may affect the interpretation of the study results or interfere with it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hematological malignancies and subjected to treatment with immune-checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence, type and severity of immune-related endocrine side effects | through study completion, an average of 2 years
  to evaluate the incidence, type and severity of immune-related endocrine side effects (thyroid disease, hypophysitis, diabetes) in patients treated with ICIs, through haematological-endocrinological management.

SECONDARY OUTCOMES:
search for predictive criteria for the appearance of immune-mediated endocrine toxicities | through study completion, an average of 2 year
  correlation between patients characteristics and occurrence of immune-mediated endocrine toxicities
impact of toxicity on the continuation of therapy | through study completion, an average of 2 year
  rate of patients who discontinued therapy due to toxicity
monitoring system for early diagnosis and management of toxicities | through study completion, an average of 2 year
  assesment of toxicities since first cycle and comparison with medical history

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No